CLINICAL TRIAL: NCT02439892
Title: Rehabilitation During Versus After Radiotherapy in Head and Neck Cancer - a Pilot Randomised Controlled Trial
Brief Title: Rehabilitation for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); LHL-Klinikkene, Røros (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDR-2012-01
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Neoplasms
Keywords: Radiotherapy; Exercise; Diet therapy; Rehabilitation; Patient Compliance; Feasibility Studies; Sample Size; Patient satisfaction
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity; Patient Compliance; Patient Satisfaction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early rehabilitation (Experimental): Exercise and nutrition during radiotherapy: Physical exercise, nutritional advice and oral nutritional supplements.
  Interventions: Behavioral: Exercise and nutrition during radiotherapy
- Late rehabilitation (Active Comparator): Multidimensional rehabilitation after radiotherapy: Physical exercise, nutritional advice, oral nutritional supplements and patient education
  Interventions: Behavioral: Multidimensional rehabilitation after radiotherapy

INTERVENTIONS:
Behavioral: Exercise and nutrition during radiotherapy — The intervention consists of physical exercise, nutritional counselling and supplements. The exercise sessions will be conducted twice a week for 30 minutes each time during the RT treatment period, and include a main part of progressive resistance training (PRT). The PRT will be conducted by conventional upper and lower body exercises at a load of 60 - 80 % of 1 repetition maximum (RM) in 3-4 sets of 6-12 repetitions. The patients will receive nutritional information and dietary advice, and up to 2 energy dense oral nutritional supplements (ONS) daily. A nutrition interview will be conducted at study baseline and individual goals and targets will be set during the first counselling and monitored during the intervention period.
  Arms: Early rehabilitation
Behavioral: Multidimensional rehabilitation after radiotherapy — The intervention consists of physical exercise, nutritional counselling and supplements and patient education. The exercise sessions will be conducted 3 times a week for 45 minutes each time during the 3 week rehabilitation programme, and include a main part of progressive resistance training (PRT). PRT will be conducted as described in the intervention during treatment. The nutritional intervention will be carried out as described in the intervention during treatment. Patient education will be run as 45-60 minutes lecture/group discussion on relevant topics, lead by health professionals.
  Arms: Late rehabilitation

SUMMARY:
Patients treated for head and neck cancer (HNC) suffer from severe side-effects such as pain and difficulties in swallowing, often leading to weight loss. More than 70 % of the weight loss is attributed to lean muscle wasting that is associated with decline in physical function, substantial fatigue and significantly decreased quality of life. Rehabilitation that includes physical exercise, nutritional counselling and oral nutritional supplements (ONS) can potentially reduce or prevent muscle wasting. The primary aim of this pilot randomised trial is to assess feasibility, evaluate patient experiences and assess preliminary effects on muscle mass, physical function, nutritional status and quality of life of rehabilitation interventions during and after radiotherapy (RT). Newly diagnosed HNC patients referred for curative RT with or without chemotherapy, will be randomised to a) rehabilitation during RT or b) rehabilitation after RT. Rehabilitation during RT will be carried out at an outpatient facility during the treatment period (6-7 weeks) and rehabilitation after RT will be carried at a rehabilitation centre and last for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell cancer (SCC) originated in the head/neck (naso, oro, hypo pharynx, larynx and oral cavity)
* Due to commence curative radiotherapy (RT) or chemoradiotherapy (CRT)
* All baseline assessments can be completed within 4 weeks prior to first cycle of RT or CRT
* Written informed consent is present
* willing to comply with study procedures

Exclusion Criteria:

* stage T1N0M0 laryngeal cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of interventions tracked by number of patients ineligible or refusing to participate, completion of interventions and attrition, adverse events and exercise/nutritional adherence. | 15 weeks

SECONDARY OUTCOMES:
Preliminary effects on skeletal muscle mass as measured by computerized tomography at lumbar vertebra 3 | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Åsmund Lund, MD PhD, Principal Investigator — St. Olavs Hospital; Stein Kaasa, prof MD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - LHL-klinikkene Røros, Røros
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Result] Sandmael JA, Bye A, Solheim TS, Stene GB, Thorsen L, Kaasa S, Lund JA, Oldervoll LM. Feasibility and preliminary effects of resistance training and nutritional supplements during versus after radiotherapy in patients with head and neck cancer: A pilot randomized trial. Cancer. 2017 Nov 15;123(22):4440-4448. doi: 10.1002/cncr.30901. Epub 2017 Jul 31. PMID 28759113
- [Result] Sandmael JA, Bye A, Solheim TS, Balstad TR, Thorsen L, Skovlund E, Kaasa S, Lund JA, Oldervoll L. Physical rehabilitation in patients with head and neck cancer: Impact on health-related quality of life and suitability of a post-treatment program. Laryngoscope Investig Otolaryngol. 2020 Mar 17;5(2):330-338. doi: 10.1002/lio2.368. eCollection 2020 Apr. PMID 32337365